CLINICAL TRIAL: NCT00239902
Title: Two-year Extension of a One-year, Multicenter, Randomized, Partially-blinded Study of the Safety and Efficacy of FTY720 Combined With Corticosteroids and Full or Reduced-dose Cyclosporine, USP [Modified] (Novartis Brand) in de Novo Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of FTY720 in de Novo Adult Renal Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720A0121E1
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Transplantation, kidney, and organ transplantation
MeSH Terms: interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study will evaluate the safety and efficacy of FTY720 combined with cyclosporine and corticosteroids in patients receiving a kidney transplant.

ELIGIBILITY:
Inclusion Criteria

- Completion of Core study

Exclusion Criteria

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 396
Dates: Start 2002-05; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB or III diagnosed by biopsy according to Banff 97 criteria within 36 months post transplant
Permanent resumption of dialysis within 36 months post transplant
Surgical removal of graft within 36 months post transplant
Death within 36 months post transplant
Discontinuation within 36 months post transplant

SECONDARY OUTCOMES:
FEV1 , FVC, DLCO within 36 months post transplant
Serum creatinine and estimated creatinine clearance within 36 months post transplant
Absolute lymphocyte count within 36 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis